CLINICAL TRIAL: NCT06149598
Title: Pain Reduction by Forced Coughing During Colposcopy Guided Cervical Biopsies: a Randomized Controlled Pilot Study
Brief Title: Coughing at Time of Cervical Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Responsible Party: Principal Investigator, Dr. med. Ziad Hilal, Principal Investigator, Zydolab - Institute of Cytology and Immune Cytochemistry
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COLPO-6
Record Dates: First submitted 2023-11-19; First posted 2023-11-29 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer; Cervical Dysplasia; Colposcopy; Pain Sensation; Cervical Biopsy
Keywords: cervical cancer; cervical dysplasia; cervical biopsy; pain; coughing; distraction
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Pain; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coughing at the time of first biopsy (Experimental): Patients are asked to cough during the first biopsy. They should not cough during the second biopsy, and no additional interventions will be performed during the second biopsy.
  Interventions: Behavioral: Coughing at the time of biopsy
- Coughing at the time of second biopsy (Active Comparator): Patients are asked to cough during the second biopsy. They should not cough during the first biopsy, and no additional interventions will be performed during the first biopsy.
  Interventions: Behavioral: Coughing at the time of biopsy

INTERVENTIONS:
Behavioral: Coughing at the time of biopsy — Patients are asked to cough or not to cough during cervical biopsy.

SUMMARY:
To investigate the effect of coughing as an intervention to reduce pain in colposcopy guided biopsy.

DETAILED DESCRIPTION:
Colposcopy is a frequently practiced examination and Colposcopy guided biopsy causes pain. A few trials Investigated whether medical interventions such as the application of lidocaine led to reduced pain perception with inconsistent results. Only one trial compared coughing versus no coughing at the moment of biopsy. Although the results of this study did not lead to a significant difference between the two study arms, coughing seems to positively affect pain perception.

Since the patients are, in the best case, their own controls when it comes to subjective parameters such as pain perception, we prefer a cross-over rather than a parallel group design.

Based on the descriptive variables for pain during biopsy with and without cough determined in the pilot study, a case estimate for a prospective randomized cross-over study will be carried out. Since two biopsies are usually taken from the cervix in daily practice, the now planned pilot study in a cross-over design envisages the following two study arms:

1. Group I: Patients cough during the first biopsy, they do not cough during the second biopsy
2. Group II: Patients cough during the second biopsy, they do not cough during the first biopsy

The primary Outcome measure is the difference in the patients' perception of pain during the first and second biopsy on the cervix (ectocervix), measured using an 11-part numerical analogue scale (11-item NAS).

ELIGIBILITY:
Inclusion Criteria:

* Completed 18 years of age
* written informed consent
* first colposcopy
* Clinically indicated colposcopy in case of an abnormal PAP smear or screening result and/or clinical abnormalities on the cervix uteri
* Necessity to take exactly two biopsies

Exclusion Criteria:

* Performing only one biopsy or more than two biopsies
* Performing an endocervical curettage (biopsy on the endocervix)
* Vaginal bleeding at the time of examination
* inadequate colposcopy
* Cervix uteri cannot be fully visualized
* Pregnancy
* Patients with insufficient German language skills
* known anxiety disorders or depressive disorders
* Treatments already carried out on the cervix uteri
* Patients with a chronic or acute illness that influences the perception of pain or lead to permanent pain due to the disease itself
* psychosomatic illnesses
* Chronic use of pain medications or psychotropic medications or other medications that may have an influence on the sensation of pain

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Difference in pain between first and second biopsy | Immediately after the examination
  the difference in the patients' perception of pain during the first and second biopsy on the cervix (ectocervix), measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.

SECONDARY OUTCOMES:
Pain perception before examination | Immediately before the start of the examination
  the patients' perception of pain before examination, measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.
Pain perception when inserting the specula | Immediately after the insertion of the specula
  the patients' perception of pain at the moment of the insertion of the specula, measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.
Pain perception when using acetic acid | Immediately after the application of acetic acid
  the patients' perception of pain at the moment of the application of acetic acid, measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.
Pain perception at first biopsy | Immediately after the first biopsy was performed
  the patients' perception of pain during the first biopsy, measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.
Pain perception at second biopsy | Immediately after the second biopsy was performed
  the patients' perception of pain during the second biopsy, measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.
Pain perception just after examination | Immediately after the removal of the specula
  the patients' perception of pain just after finishing the examination, measured using an 11-part numerical analogue scale (11-item NAS). The numerical analogue scale consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (score 0) and 'pain as bad as it could be' (score 10). Women will be asked to mark her pain level on the line between the two endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Zydolab - Institute of Cytology and Immune Cytochemistry, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No